CLINICAL TRIAL: NCT07018557
Title: Impact of Eszopiclone on Blood Pressure in Patients With Insomnia and Hypertension (PRYSMA-HTN)
Acronym: PRYSMA-HTN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Associate Professor of Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73710523.3.0000.0068; Investigator initiated Study (Other: Heart Institute (InCor), University of Sao Paulo Medical School, Brazil)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Insomnia; Hypertension
Keywords: Insomnia; Hypertension; Blood Pressure; Treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hypertension | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo + sleep hygiene (Placebo Comparator): Placebo pill (identical to the active treatment) + sleep counseling for improving insomnia
  Interventions: Drug: Placebo
- Eszopiclone + sleep hygiene (Active Comparator): Active treatment for insomnia + sleep counseling
  Interventions: Drug: Eszopiclone 3 mg

INTERVENTIONS:
Drug: Eszopiclone 3 mg — Eszopiclone is an FDA-approved treatment for insomnia in those who have difficulty falling asleep and for patients with difficulty staying asleep (sleep maintenance).
  Arms: Eszopiclone + sleep hygiene
Drug: Placebo — Placebo pills identical to the active comparator.
  Arms: Placebo + sleep hygiene

SUMMARY:
Insomnia is a common sleep disorder characterized by difficulty falling asleep, staying asleep, or both, despite appropriate opportunities for getting sleep. Growing evidence has associated insomnia with prevalent and incidence of hypertension. However, the impact of the pharmacologic treatment of insomnia on office blood pressure (BP) and 24-h ambulatory BP monitoring (ABPM) in unclear. Therefore, the aim of this study is to evaluate the impact of eszopiclone, a non-benzodiazepine hypnotic that binds to certain subunits of the gamma-aminobutyric acid type A receptors GABA-A (such as α1, α3, and α5) promoting relaxation and sleep. Eszopiclone is an FDA-approved treatment for insomnia in those who have difficulty falling asleep and for patients with difficulty staying asleep (sleep maintenance).

DETAILED DESCRIPTION:
We will consecutively evaluate the presence of insomnia in adult patients with hypertension under regular treatment recruited from the outpatient clinic at the Heart Institute (InCor).

The following exams will be made:

1. Definition of the presence of insomnia following the criteria from DSM V and severity by the insomnia severity index.
2. Evaluation of the Pittsburgh Sleep Quality Index.
3. Evaluation of daytime sleepiness by the Epworth Sleepiness Scale.
4. Evaluation of anxiety disorder by the Generalized Anxiety Disorder (GAD-7)
5. Beck form for depression evaluation.
6. Detection of sleep apnea using a portable monitor (BiologixTM) Patients that fulfilled the inclusion criteria will be submitted to a 1-month run-in period before randomization with pill counting for improving medical adherence and defining baseline BP. Then patients with be randomized to sleep hygiene + eszopiclone or sleep hygiene + placebo for 3 months (double-blind study design). We will collect demographic and anthropometric data, as well as concomitant comorbidities, medications, standard BP measurements (office and ABPM) at baseline and after 3 -months.

The main hypothesis is that pharmacological treatment, as compared to placebo, will be able to improve insomnia in parallel to a significant decrease in 24-h ABPM (primary outcome). We will also evaluate absolute decrease of daytime and nighttime BP, % of 24-h, daytime, and nighttime BP control, % non-dipping BP, office BP, sleep quality and improvement in insomnia severity index scale as secondary outcomes. Exploratory analysis evaluating the effects of eszopiclone according to the type of insomnia (initial or sleep-onset insomnia, middle or maintenance insomnia and terminal or late insomnia). We also explored whether the results will be influenced by the presence of untreated sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Adults (30 to 75 years-old)
* BMI <40Kg/m2;
* Availability to participate
* History of HBP under regular treatment (systolic pressure between 130-160 and diastolic pressure between 80-100 mmHg).

Exclusion Criteria:

* Use of benzodiazepines or "Z" drugs;
* Night workers;
* History of severe chronic obstructive pulmonary disease (COPD);
* Heart failure (ejection fraction <40% on echocardiogram);
* Prior stroke;
* Generalized anxiety disorder (GAD-7 >14 points) and severe depression (Beck);
* Severe liver disease;
* Alcohol abuse;
* Advanced chronic kidney disease 4 or 5 (glomerular filtration rate <30ml/min/1.73m2);
* Patient who is on loop diuretics;
* Patient with type 1 diabetes;
* Patient with decompensated type 2 diabetes (Glycated hemoglobin >10%);
* Urinuria Incontinence;
* Prostatism;
* History of active cancer;
* Pregnancy;
* Complex sleep behaviors, suicidal behavior.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of insomnia treatment on blood pressure (evaluated by Ambulatory blood pressure monitoring) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on 24-h blood pressure by ABPM (mmHg).

SECONDARY OUTCOMES:
Efficacy of insomnia treatment on daytime and nighttime blood pressure (evaluated by Ambulatory blood pressure monitoring) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on daytime and nighttime blood pressure BP (mmHg).
Efficacy of insomnia treatment on 24-h, daytime, and nighttime BP control (evaluated by Ambulatory blood pressure monitoring) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on 24-h, daytime, and nighttime BP control (%).
Efficacy of insomnia treatment on non-dipping BP pattern (evaluated by Ambulatory blood pressure monitoring) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on non-dipping BP (%).
Efficacy of insomnia treatment on blood pressure (evaluated by office blood pressure) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on office BP (mmHg).
Efficacy of insomnia treatment on sleep quality (evaluated by Pittsburgh Sleep Quality Index) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on sleep quality (absolute values).
Efficacy of insomnia treatment on insomnia severity (evaluated by insomnia severity index) | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on insomnia severity (absolute values).

OTHER OUTCOMES:
Efficacy of insomnia treatment on blood pressure based on the type of insomnia | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on blood pressure according to the type of insomnia (initial or sleep-onset insomnia, middle or maintenance insomnia and terminal or late insomnia).
Efficacy of insomnia treatment on blood pressure according to sleep apnea status | 3 months
  To assess the impact of treatment of insomnia with eszopiclone on blood pressure in patients with and without sleep apnea.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano F. Drager, MD, PhD, Study Chair — University of Sao Paulo Medical School
Locations (1):
- Academic Research Organization - Heart Institute (InCor), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided